CLINICAL TRIAL: NCT06800300
Title: Identification of the Risk of Remote Pulmonary Hypertension in Preterm Births.
Acronym: Iper-NeoRisk
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Iper-NeoRisk
Record Dates: First submitted 2025-01-09; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: PreTerm Neonate; Pulmonary Hypertension of Newborn; Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to learn about the prevalence of pulmonary hypertension and right ventricular dysfunction in patients born prematurely, at birth and at a distance, and the association with the development of pulmonary bronchodysplasia, so that screening programs can be set up in the future and proper treatment can be initiated in a timely manner.

DETAILED DESCRIPTION:
This study aims to learn about the prevalence of pulmonary hypertension and right ventricular dysfunction in patients born prematurely, at birth and at a distance, and the association with the development of pulmonary bronchodysplasia, so that screening programs can be set up in the future and proper treatment can be initiated in a timely manner. Enrolled patients, should asymptomatic pulmonary hypertension be diagnosed, will be able to be taken to dedicated outpatient clinics and initiate appropriate treatment if indicated. The primary goal of this study is to evaluate the incidence of late pulmonary arterial hypertension and/or right ventricular dysfunction in a cohort of former preterm patients. The study will also provide a greater awareness of the epidemiology of pulmonary hypertension and right ventricular dysfunction in these patients and allow appropriate screening and follow-up to be planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with prematurity with gestational age less than 30 weeks evaluated at outpatient clinics dedicated to neonatal follow-up of participating health care providers during the study data collection period.
* Obtaining informed consent.

Exclusion Criteria:

* Prenatal or postnatal diagnosis of genetic disease;
* Concomitant presence of congenital heart disease except interatrial defect or patency of the ductus arteriosus;
* Concomitant presence of diaphragmatic hernia

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants of gestational age (EG) ≤30 weeks, at birth and/or during neonatal follow-up afferent to the Neonatology Operating Units participating in the study (Operating Unit of Neonatology at the Policlinico Sant'Orsola Malpighi Hospital in Bologna, Italy, and the Complex Operating Unit of Neonatology at the Policlinico Agostino Gemelli Hospital in Rome, Italy.)
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Identify the incidence of pulmonary hypertension or right ventricular dysfunction in patients born prematurely at a 1-year follow-up. | From enrollment to the 1 year follow up
  Identify the prevalence of pulmonary hypertension and right ventricular dysfunction in patients born prematurely

SECONDARY OUTCOMES:
to define risk classes for the development of pulmonary arterial hypertension in patients born prematurely. | From enrollment to the 1 year follow up
  Echocardiographic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Donti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO
  - Policlinico Agostino Gemelli di Roma, Roma, RM